CLINICAL TRIAL: NCT03180099
Title: Efficiency of Thoracolumbar Interfascial Plane Block in Lumbar Disk Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erzurum Palandöken State Hospital (Other Government)
Responsible Party: Principal Investigator, Erkan Cem ÇELİK, Consult of Anesthesiologhy, Erzurum Palandöken State Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ErzurumPSH
Record Dates: First submitted 2017-04-29; First posted 2017-06-08 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Pain
Keywords: Lumbar Disk Hernia; Thoracolumbar Interfascial Plane Block; Lumbar Disk Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Anesthesia, Epidural

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thoracolumbar Interfascial Plane Block (Active Comparator): Bilateral ultrasound guided thoracolumbar interfascial plane block
  Interventions: Drug: Bupivacaine
- Epidural Block (Active Comparator): Epidural Block
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Ultrasonically assisted, 0.5-1 mL 0.9% NaCl test is given between m.longissimus and m.iliocostalis to confirm the position of the needle and local anesthetic drugs will be given here
  Other Names: Thoracolumbar Interfascial Plane Block
  Arms: Thoracolumbar Interfascial Plane Block
Drug: Bupivacaine — 20 ml %0.1 Bupivacaine administered to Epidural Space
  Other Names: Epidural Block
  Arms: Epidural Block

SUMMARY:
Objectives:Lomber disc hernia is one of the most common diseases in Turkey. The prevalence in various studies is between 60-80% and incidence is between 1-3% for the entire population,Goal of TLIP is to provide a same impact in the thoracolumbar region, like thoracoabdominal plane block (TAP) diminish the pain in the abdominal surgery Methods: The study design was approved by the locale ethics committee. This double-blinded, randomized, controlled clinical trial recruited 50 patients who were candidated for surgical operations on lumbar disc hernia surgery. . Patients will be divided into two groups as Group T (TLIP block) and Group E (Epidural group).In group T, TLIP block will be applied before anesthesia and surgery and evaluate block efficiency with temperature discrimination and pin-prick test. During the TLIP block, block fluid will have total volume of 20 mL of 0.5% bupivacaine.). In Group E, after surgery, total of 20 ml of 0.1% bupivacaine and 50 mcg of fentanyl will be performed in the epidural space with direct vision by the surgeon.For the postoperative analgesia, patient controlled analgesia device will be administered as 20 mg/h continue dose tramadol and administered 10 mg bolus dose tramadol if patient need a rescue dose. Nausea-vomiting, tramadol consumption, bolus dose intervention and visual analog scale value in the postoperative 0-4., 4-12., and 12-24. hour interval will be assess and results will be record.

DETAILED DESCRIPTION:
Efficiency of Thoracolumbar Interfascial Plane Block in Lumbar Disk Surgery Lomber disc hernia is one of the most common diseases in Turkey. The prevalence in various studies is between 60-80% and incidence is between 1-3% for the entire population, If adequate analgesia isn't achieved in postoperative period, the patients can faced with postoperative pain due to lomber disc hernia. In fact, as a result of inadequate analgesia chronic pain can be develop, and patients can be suffered by this pain for long years Thoracolumbar interfascial blok, was defined by Hand et al, descibed for reduce pain of thoracolumbar region surgery. After afferent fibers separate from medulla spinalis, they're called r.anterior and r.posterior. While r. anterior spreads to anterior abdominal wall, r.posterior spreads to thoracolumbar region. Goal of TLIP is to provide a same impact in the thoracolumbar region, like thoracoabdominal plane block (TAP) diminish the pain in the abdominal surgery.

The study design was approved by the locale ethics committee. This double-blinded, randomized, controlled clinical trial recruited 50 patients aged between 18 and 65 years with the American society of anesthesiologists (ASA) physical status classification systems I/II who were candidated for surgical operations on lumbar disc hernia surgery. All the participants will be asked to sign an informed consent form after having been provided with details of the aim and proceedings of the study. Patients will excluded from the study if they have a neurological and neuromuscular disorders, psychiatric problems, cardiopulmoner diseases, coagulopathy, infections or allergy to local anesthetic agents. Patients will be divided into two groups as Group T (TLIP block) and Group E (Epidural group).

Prior to the study, a power analysis was performed to determine the necessary number of patients in each group. With a two-sided type I error of 5% and study power at 80%, it was estimated that 25 patients would be needed in each group 20 gauge cannulas are placed over the left hand of the patient in the operating room and 4 ml kg-1% 0.9% NaCl infusion will be made. The age, weight and sex of the patients will record and the ECG, SpO2, non-invasive blood pressure monitor will be used as standard in the operating room. Routine anesthesia induction in both groups will be performed with 2 mg kg-1 propofol 50 mcg fentanyl and 0.6 mg kg-1 rocuronium anesthesia with 40/60% O2 / N2O 2% sevofloran.

In group T, TLIP block will be applied before anesthesia and surgery and evaluate block efficiency with temperature discrimination and pin-prick test. During the TLIP block, block fluid will have total volume of 20 mL of 0.5% bupivacaine. TLIP block implementation will be made in accordance with the asepsis antisepsis rules. Ultrasonically assisted, 0.5-1 mL 0.9% NaCl test is given between m.longissimus and m.iliocostalis to confirm the position of the needle and local anesthetic drugs will be given here (according to new approach). In Group E, after surgery, total of 20 ml of 0.1% bupivacaine and 50 mcg of fentanyl will be performed in the epidural space with direct vision by the surgeon. After, patients will be administered with 0,01 mg kg atropine iv and 0,02 mg kg neostigmine iv and extubated at the end of the surgery, they will be taken to PACU. For the postoperative analgesia, patient controlled analgesia device will be administered as 20 mg/h continue dose tramadol and administered 10 mg bolus dose tramadol if patient need a rescue dose. Nausea-vomiting, tramadol consumption, bolus dose intervention and visual analog scale value in the postoperative 0-4., 4-12., and 12-24. hour interval will be assess and results will be record.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 70 years with the American society of anesthesiologists (ASA) physical status classification systems I/II who were candidated for surgical operations on lumbar disc hernia surgery

Exclusion Criteria:

* have a neurological and neuromuscular disorders, psychiatric problems, cardiopulmoner diseases, coagulopathy, infections or allergy to local anesthetic agents.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-10 (Estimated); Primary Completion 2017-11-11 (Estimated); Study Completion 2017-12-11 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption | [Time Frame: First 24 hours total opioid consumption]
  First 24 hours total fentanyl consumption with patient controlled analgesia

SECONDARY OUTCOMES:
Visual Analogue Pain Score | [Time Frame: postoperative first hour]
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at first hour postoperatively
Visual Analogue Pain Score | [Time Frame: postoperative second hour]
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at second hour postoperatively.
Visual Analogue Pain Score | [Time Frame: postoperative 4th hour]
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 4th hour postoperatively
Visual analog pain score | [Time Frame: postoperative 8th hour]
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 8th hour postoperatively
Visual analog pain score | [Time Frame: postoperative 12th hour]
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 12th hour postoperatively.
Visual analog pain score | [Time Frame: postoperative 24th hour]
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 24th hour postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Erkan Cem ÇELİK, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Hand WR, Taylor JM, Harvey NR, Epperson TI, Gunselman RJ, Bolin ED, Whiteley J. Thoracolumbar interfascial plane (TLIP) block: a pilot study in volunteers. Can J Anaesth. 2015 Nov;62(11):1196-200. doi: 10.1007/s12630-015-0431-y. Epub 2015 Jul 7. PMID 26149600
- [Result] Ahiskalioglu A, Alici HA, Selvitopi K, Yayik AM. Ultrasonography-guided modified thoracolumbar interfascial plane block: a new approach. Can J Anaesth. 2017 Jul;64(7):775-776. doi: 10.1007/s12630-017-0851-y. Epub 2017 Feb 27. No abstract available. PMID 28243853